CLINICAL TRIAL: NCT03375827
Title: Feasibility of an Individualized Goals of Care Discussion Guide for Advanced Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Jeffrey Peppercorn, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-398
Record Dates: First submitted 2017-11-06; First posted 2017-12-18 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survey QOL (Experimental): * Study participants will be provided with the Individualized Goals of Care Discussion Guide (IGCDG) consisting of a brief pamphlet and the IGCDG questionnaire.
  * Participants will be asked to complete the IGCDG questionnaire prior to their next visit.
  * Participants will also complete an 8-week follow-up survey after the clinic visit to evaluate the impact on patient satisfaction with care, communication, and care received.
  Interventions: Other: IGCDG

INTERVENTIONS:
Other: IGCDG — The IGCDG reviews topics of concern for patients with metastatic breast cancer.

SUMMARY:
This research study is evaluating whether asking patients to fill out a brief survey about their goals and preferences for care and giving this survey to their clinician before the next visit helps improve communication and decision-making in breast cancer care.

DETAILED DESCRIPTION:
The purpose of this study is to understand patient preferences for communication and decision-making for advanced breast cancer. The investigators want to better understand what topics the participant wants their doctors and nurses to address with the participant in clinic, and the investigators want to evaluate whether asking patients to fill out a brief survey about their goals and preferences for care and giving this survey to their clinician before the next visit is a good idea that helps to improve communication and decision-making in breast cancer care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Diagnosed with stage IV breast cancer within the past 3 years
* Receiving care at the MGH Cancer Center
* Verbal and written fluency in English
* Within 6 weeks of a new line of breast cancer therapy and/or progression on scans and/or a change in current breast cancer therapy regimen

Exclusion Criteria:

* Unwilling or unable to participate in the study
* Is medically or otherwise unable to participate (as determined by a physician or study PI)
* Enrolled in hospice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 2 years
  The investigators will evaluate the primary hypothesis, that administration of the IGCDG in a breast oncology clinic is feasible, by evaluating the recruitment rate. Recruitment will be calculated as the number of patients who choose to participate divided by the number approached to enroll. A recruitment rate of greater than 50% will be deemed feasible. Each of the 3 distinct components of feasibility (recruitment rate, attrition rate, and change in distress) must be met for the administration of the Individualized Goals of Care Discussion Guide to be deemed feasible.
Attrition rate | 2 years
  The investigators will evaluate the primary hypothesis, that administration of the IGCDG in a breast oncology clinic is feasible, by evaluating the attrition rate. Attrition will be calculated as the number of participants who to do not complete the follow-up survey divided by the number enrolled. An attrition rate of less than 32% will be deemed feasible. Each of the 3 distinct components of feasibility (recruitment rate, attrition rate, and change in distress) must be met for the administration of the Individualized Goals of Care Discussion Guide to be deemed feasible.
Change in distress | 8 weeks after the IGCDG was provided to participant's clinician
  The investigators will evaluate the primary hypothesis, that administration of the IGCDG in a breast oncology clinic is feasible, by evaluating the change in distress as measured by the NCCN distress thermometer between baseline administration and the 8-week follow-up survey. Lack of detection of a significant increase between baseline and follow-up distress scores among the participants will be interpreted as supporting feasibility. A significant increase in distress will be defined as >50% of participants having an increase in distress ≥3 between baseline and follow-up. Each of the 3 distinct components of feasibility (recruitment rate, attrition rate, and change in distress) must be met for the administration of the Individualized Goals of Care Discussion Guide to be deemed feasible.

SECONDARY OUTCOMES:
Evaluate baseline preferences for care among patients with metastatic breast cancer via the Individualized Goals of Care Discussion Guide (IGCDG) questionnaire | baseline
  The IGCDG questionnaire reviews topics of concern for patients with metastatic breast cancer, such as goals of cancer treatment and priorities for discussions with the patient's clinician. This is a descriptive, study specific measure.
The Satisfaction with Decision Making Scale | 8 weeks after the IGCDG was provided to participant's clinician
  This is a six item validated scale designed to measure patient satisfaction with medical decision making. Participants rate their level of agreement on a 5-point scale with statements regarding medical decision-making. (1 = strongly agree; 5 = strongly disagree) . Lower scores indicate higher inclusion of the patient in decision-making.
The Decisional Conflict Scale | 8 weeks after the IGCDG was provided to participant's clinician
  This is a 16-item Likert scale with proven validity and reliability. Scores range from 1 to 5, with higher scores suggesting increased difficulty and conflict over decision making.
Modified Control Preferences Scale | 8 weeks after the IGCDG was provided to participant's clinician
  This 2 question scale is used to measure a participant's desired and actual participation in decision-making. As in prior work, the investigators have collapsed responses into 3 choices: decisions are made mainly by the patient, decisions are made equally, and decisions are made mainly by the clinician. Analysis is based on comparison of the participants reported desired role in decision making and actual role, with greater concordance indicating decision making that is aligned with the participants preferences.
Patient Satisfaction with Cancer Care | 8 weeks after the IGCDG was provided to participant's clinician
  The Patient Satisfaction with Cancer Care measure is a validated 18 item tool with responses on a 5 point Likert scale designed specifically to assess satisfaction among patients from diverse socio-demographic backgrounds. The investigators have modified the scale to remove 3 questions that were not relevant for this study population. Total score for this scale is calculated by adding all component scores, with lower scores indicating higher satisfaction with care.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Peppercorn, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No